CLINICAL TRIAL: NCT03921632
Title: Impact of an Oral Health Intervention Among a Group of Patients With Eating Disorders (Anorexia Nervosa and Bulimia Nervosa)
Brief Title: Impact of an Oral Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: 15-3295
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Eating Disorder
Keywords: Anorexia nervosa; Bulimia
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Education Program Effectiveness (Experimental): Outpatients and inpatients from UNC Center of Excellence for Eating Disorders clinic
  Interventions: Behavioral: Smiles Matter Oral Health Education Series

INTERVENTIONS:
Behavioral: Smiles Matter Oral Health Education Series — Three sessions scheduled 2 weeks apart consisting of 15-20 minutes of didactic learning, 10 minutes of a group/personal exercise, and 10 minutes of questions that the patients have on the topic discussed that day

SUMMARY:
This pilot study will assess the effectiveness of an original oral health education program on affecting the behaviors of patients diagnosed with eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the UNC Center for Excellence for Eating Disorders inpatient unit or outpatient clinic.
* Diagnosis of anorexia nervosa or bulimia nervosa
* Aged 13-50 years
* English-speaking

Exclusion Criteria:

* Decisionally impaired (i.e., Incapable of providing informed consent in the opinion of the primary care provider in UNC Center for Excellence for Eating Disorders)
* Involuntarily committed to the inpatient service of the UNC Department of Psychiatry

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Percent Change of Participants Able to Correctly Identify Possible Oral Effects of Eating Disorders | Baseline, Week 6
  A multiple choice survey inquiring about potential effects of eating disorders (e.g., Tooth erosion, Probable erosion sites, Tooth sensitivity, Dry mouth, Enlarged saliva glands, Oral cancer, or No pain) and Positive Self-Perception (e.g., Confidence, Appearance, Kissing, General Health Attendance) posed as Yes/No response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roberts, DDS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Center of Excellence for Eating Disorders Clinic, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared.
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Silverstein LS, Haggerty C, Sams L, Phillips C, Roberts MW. Impact of an oral health education intervention among a group of patients with eating disorders (anorexia nervosa and bulimia nervosa). J Eat Disord. 2019 Sep 5;7:29. doi: 10.1186/s40337-019-0259-x. eCollection 2019. PMID 31508232